CLINICAL TRIAL: NCT04090749
Title: Caregiver Support in the Context of Multiple Chronic Conditions: Randomized Waitlist Control Trial
Brief Title: Caregiver Support in the Context of Multiple Chronic Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB00203584; 5P30NR018093 (NIH)
Record Dates: First submitted 2019-09-12; First posted 2019-09-16 (Actual); Results first posted 2023-12-22 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Caregiver Burnout
Keywords: coping; resilience; quality of life
MeSH Terms: conditions — Caregiver Burden

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The research assistant collecting data will be blinded to group assignment for each participant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Open Label Group (Experimental): In this arm, 5 participants will be enrolled in the intervention without blinding or randomization. The intervention and study delivery will be improved based on findings from this arm.
  Interventions: Behavioral: Caregiver-Support
- Waitlist Control (Other): The waitlist control group (n=20) will be provided written materials with community resources for caregivers during the first 16 weeks, then the intervention will begin.
  Interventions: Behavioral: Caregiver-Support
- Immediate Intervention (Experimental): The immediate intervention group (n=20) will receive the intervention during weeks 0-16. There will be assessment at week 32 to examine maintenance on primary and secondary outcomes.
  Interventions: Behavioral: Caregiver-Support

INTERVENTIONS:
Behavioral: Caregiver-Support — intervention incorporating 5 individualized, nurse-led, home-based sessions, with telephone check-ins and text reminders, according to participant preference. Caregiver-Support will help caregivers articulate statements of purpose in life, set goals to address fatigue and caregiver burden, provide instrumental support through a benefits check up and promote identification and increased connection with the caregiver's social network.

SUMMARY:
This research is being done to learn whether services to the caregiver to provide emotional, instrumental and social support can improve quality of life and other outcomes. The Caregiver-Support program provides services that are not usually available to caregivers of persons with heart failure and other chronic conditions.

DETAILED DESCRIPTION:
Family caregivers who care for older adults living with multiple chronic conditions, including heart failure (HF), provide substantial cost savings to the US healthcare system. While caregiving can be meaningful and rewarding, extensive research also demonstrates high rates of chronic disease, fatigue and physiologic measures such as stress hormones among caregivers. Family caregivers are often left juggling caregivers' loved one's healthcare as well as caregivers' own. Unmet needs have been identified including increased stress, financial strain and social isolation, but interventions to address these needs in HF caregivers have had mixed results. Due to the limited impact of many caregiver interventions, experts have called for a greater understanding of the dynamic and contextual factors of family caregiving including resources, needs and social support with an increased focus on individualization of interventions for high-risk caregivers to improve outcomes.Following a mixed methods study to better understand these contextual factors and to address this gap between the evidence and uptake of proven strategies by caregivers, the study team has developed a resilience-promoting intervention to improve quality of life for family caregivers of individuals with multiple chronic conditions, including HF, Caregiver-Support. Caregiver-Support will help caregivers articulate statements of purpose in life, set goals to address fatigue and caregiver burden, provide instrumental support through a benefits check up and promote identification and increased connection with the caregiver's social network.

The first phase of the study will be an open label pilot (N=5) followed by a single-masked, two-group, randomized trial (N=40) to test the feasibility and gauge an initial effect size of the intervention. Participants will be visited by study staff in participants' homes for all data collection and intervention visits. Participants will be randomized to receive either the immediate intervention group or the waitlist control group. In the waitlist control group, participants will receive usual care for the first 16 weeks (which is limited to printed materials provided in the clinic) and then begin the intervention.

The intervention will consist of 5 in-home sessions with a nurse interventionist. Each participant will receive each intervention component but interventionists will systematically tailor content to the participants' goals based on protocols. All participants will be reassessed at 16 weeks (in person) and 32 weeks (by phone) by a research assistant (RA) masked to treatment condition. The primary outcome will be improvement in quality of life between baseline and 16 weeks. Other endpoints include group differences in fatigue, caregiver burden, self-reported and physiological measures of resilience up through 32 weeks after the intervention. The investigators will also examine the acceptability of the intervention using intervention compliance and participant satisfaction data.

ELIGIBILITY:
Inclusion Criteria:

* Primary family caregivers, will be identified by patients and providers in the Bridge Clinic
* must live with the patient or visit at least 3 times per week for the purposes of care provision
* provide support for at least one Instrumental Activity of Daily Living,
* Be able to speak English.

Exclusion Criteria:

* Caregivers with terminal diagnosis will be excluded as goal-setting at end of life may be different than without a terminal diagnosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2020-08-28 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martha Abshire, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins School of Nursing, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Background] Abshire Saylor M, Pavlovic NV, DeGroot L, Jajodia A, Hladek MD, Perrin N, Wolff J, Davidson PM, Szanton S. Strengths-building through life purpose, self-care goal setting and social support: Study protocol for Caregiver Support. Contemp Clin Trials Commun. 2022 May 5;28:100917. doi: 10.1016/j.conctc.2022.100917. eCollection 2022 Aug. PMID 35602009
- [Result] Abshire Saylor M, Pavlovic N, DeGroot L, Peeler A, Nelson KE, Perrin N, Gilotra NA, Wolff JL, Davidson PM, Szanton SL. Feasibility of a Multi-Component Strengths-Building Intervention for Caregivers of Persons With Heart Failure. J Appl Gerontol. 2023 Dec;42(12):2371-2382. doi: 10.1177/07334648231191595. Epub 2023 Sep 14. PMID 37707361

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 38 enrolled participants, 3 withdrew and 8 were lost to follow up prior to baseline data collection and randomization.
Groups:
- Open Label Pilot: This group was the first consented participants and was not randomized, but instead all participants received the intervention. Information from this group was used to test study procedures and make final minor changes to the intervention protocol.
Period: Open Label Pilot
Arm/Group | Open Label Pilot | Immediate Intervention | Waitlist Control
Started | 3 | 0 | 0
Completed | 2 | 0 | 0
Not Completed | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Period: Pilot Trial
Arm/Group | Open Label Pilot | Immediate Intervention | Waitlist Control
Started | 0 | 12 | 12
Completed | 0 | 10 | 11
Not Completed | 0 | 2 | 1
Not completed — Care recipient of enrolled caregiver died | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Immediate Intervention: The immediate intervention group received the intervention during weeks 0-16. There was an assessment at week 32 to examine maintenance on primary and secondary outcomes.
  Caregiver-Support: intervention incorporating 5 individualized, nurse-led, home-based sessions, with telephone check-ins and text reminders, according to participant preference. Caregiver-Support will help caregivers articulate statements of purpose in life, set goals to address fatigue and caregiver burden, provide instrumental support through a benefits check up and promote identification and increased connection with the caregiver's social network.
- Waitlist Control: The waitlist control group was provided written materials with community resources for caregivers during the first 16 weeks, then the intervention began.
- Total: Total of all reporting groups
Arm/Group | Open Label Pilot | Immediate Intervention | Waitlist Control | Total
Number analyzed (Participants) | 3 | 12 | 12 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (12) | 55.8 (19.6) | 62.1 (13.9) | 59 (16.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 11 | 11 | 25
  Male | 0 | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 7 | 1 | 10
  White | 1 | 5 | 11 | 17
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 12 | 12 | 27
Caregiver Burden [Mean (Standard Deviation); unit: units on a scale] — The Zarit Caregiver Burden Interview is a 12 item measure with higher scores representing higher feelings of burden; the range of summed scores is 0-48.
  units on a scale | 14.8 (10) | 15.1 (11.2) | 14.4 (15.3) | 14.75 (12)
Quality of Life (mental) [Mean (Standard Deviation); unit: units on a scale] — The Short Form Health Survey (36 items) measures self-rated quality of life using 8 sub-scales. Items are scored on a 0-100 range, with total scores averaged for each subscale. The mental health component is an average of 4 sub-scale scores. Higher scores indicate a more favorable health state.
  units on a scale | 65.2 (17.1) | 63.4 (18.8) | 77.6 (20.1) | 70.5 (19.5)

OUTCOME MEASURES:

1. Primary Outcome: Quality of Life as Assessed by the Short Form Health Survey
Description: The Short Form Health Survey (36 items) measures self-rated quality of life using 8 sub-scales. Items are scored on a 0-100 range, with total scores averaged for each subscale. The eight domains are also averaged to create an overall score from 0-100. Higher scores indicate a more favorable health state.
Time Frame: 16 weeks and 32 weeks
Population: 1 open label pilot participant did not start the intervention after completing the baseline surveys and did not complete subsequent timepoints for the surveys. The open label pilot participants did not complete the 32 week data collection.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open Label Pilot | Immediate Intervention | Waitlist Control
Number analyzed (Participants) | 2 | 10 | 11
units on a scale
  16 weeks | 72.3 (25.9) | 74.1 (20.6) | 70.4 (20.6)
  32 weeks: number analyzed (Participants) | 0 | 10 | 11
  32 weeks |  | 76.1 (21.2) | 74.0 (21.2)

2. Secondary Outcome: Fatigue as Assessed by the Patient-Reported Outcomes Measurement Information System (PROMIS)
Description: The PROMIS 7-item fatigue measure has a score range from 0-35 with higher scores indicating higher levels of fatigue. We use T-scores for analysis (where standard scores with a mean of 50 and standard deviation of 10 in the U.S. general population).
Time Frame: 16 weeks and 32 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open Label Pilot | Immediate Intervention | Waitlist Control
Number analyzed (Participants) | 2 | 10 | 11
units on a scale
  16 weeks | 50.3 (8.1) | 54.3 (7.7) | 49.1 (10.7)
  32 weeks: number analyzed (Participants) | 0 | 10 | 11
  32 weeks |  | 48.2 (9) | 53.6 (14.9)

3. Secondary Outcome: Caregiver Burden as Assessed by the Oberst Caregiving Burden Scale
Description: The investigators will use the task difficulty and time caring subscales of the Oberst Caregiving Burden Scale, which include 15 likert scale items. Scores range from 15-75. Higher scores indicate greater task difficulty and more time spent on each task, higher burden.
Time Frame: 16 weeks and 32 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open Label Pilot | Immediate Intervention | Waitlist Control
Number analyzed (Participants) | 2 | 10 | 11
units on a scale
  16 weeks | 44 (4.8) | 46 (3.4) | 39.3 (4.5)
  32 weeks: number analyzed (Participants) | 0 | 10 | 11
  32 weeks |  | 38.5 (3.2) | 37.5 (4.6)

4. Secondary Outcome: Caregiver Burden as Assessed by the Zarit Caregiver Burden Interview (ZBI)
Description: The ZBI is a 12 item measure with higher scores representing higher feelings of burden; the range of summed scores is 0-48.
Time Frame: 16 weeks and 32 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open Label Pilot | Immediate Intervention | Waitlist Control
Number analyzed (Participants) | 2 | 10 | 11
units on a scale
  16 weeks | 13.9 (10.2) | 11.3 (10.6) | 14.8 (10.6)
  32 weeks: number analyzed (Participants) | 0 | 10 | 11
  32 weeks |  | 10.2 (9) | 9.9 (9)

5. Other Pre Specified Outcome: Change in Interleukin 6 (ng/mL)
Description: Participants will wear a non-occlusive sweatpatch to collect interleukin 6. Higher levels of interleukin 6 suggest increased activation of inflammatory response and decreased resilience to stress.
Time Frame: Baseline, 16 weeks and 32 weeks
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Change in Interleukin 10 (pg/ml)
Description: Participants will wear a non-occlusive sweatpatch to collect interleukin 10. Higher levels of interleukin 10 suggest increased activation of the anti-inflammatory response and increased resilience to stress.
Time Frame: Baseline, 16 weeks and 32 weeks
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Change in Resilience to Stress as Assessed by Heart Rate Variability
Description: Participants will touch a finger pad for 2-5 minutes to obtain heart rate variability. Heart rate variability is assessed through multiple calculations including: percentage of pairs of adjacent N-N intervals differing by more than 50 milliseconds (pNN50), high-frequency power (HF power), and low frequency to high frequency (LF/HF) ratio. Higher pNN50, HF power and LF/HF ratio levels suggest increased resilience to stress.
Time Frame: Baseline, 16 weeks and 32 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 32 weeks
Description: We used the clinicaltrials.gov definition of adverse reporting
Arm/Group | Waitlist Control | Immediate Intervention | Open Label Pilot
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/3
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-29): https://cdn.clinicaltrials.gov/large-docs/49/NCT04090749/Prot_SAP_000.pdf